CLINICAL TRIAL: NCT05872737
Title: Facilitator-guided Acceptance and Commitment Bibliotherapy for Parents of Young Children With Neurodevelopmental Disorders: A Randomised Controlled Trial
Brief Title: FAB Programme for Parents of Children With NDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Sheng Kung Hui Welfare Council Limited (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTEC-2022-0091
Record Dates: First submitted 2023-05-04; First posted 2023-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Neurodevelopmental Disorders; Intellectual Disability; Specific Learning Disorder; Communication Disorders; Motor Disorders
Keywords: Neurodevelopmental disorders; Facilitator-guided Acceptance and Commitment Bibliotherapy; Parental psychological health; Parenting stress; Repeated-measures parallel-group design; Randomized controlled trial; Psychological flexibility; Hong Kong; Acceptance and Commitment Therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Intellectual Disability; Specific Learning Disorder; Communication Disorders; Motor Disorders | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: A multi-centre, two-arm randomised controlled trial (RCT) with a repeated-measures parallel-group design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB) (Experimental): A 12-week facilitator-guided Acceptance and Commitment Bibliotherapy, which includes general parenting advice and is delivered via a website
  Interventions: Behavioral: Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB)
- Control Group (Placebo Comparator): Routine family support services and four video-conferencing sessions over the course of 12 weeks
  Interventions: Behavioral: General Parenting Education and Advice

INTERVENTIONS:
Behavioral: Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB) — The Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB) is a 12-week self-help parenting program that integrates Acceptance and Commitment Therapy (ACT) principles with web-based modules and group-based sessions. The program includes a self-help workbook/manual and ACT protocols that cover various self-help exercises such as guided imagery, grounding, mindfulness, and values clarifications. To make the programme more relatable to Hong Kong parents caring for children with NDD, storytelling vignettes and therapeutic narratives will be included. Parents will work on each module at their own pace within 2-3 weeks and meet with trained facilitators in a video-conferencing format after completing each module to review their progress and learn positive parenting techniques.
  Other Names: FAB
  Arms: Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB)
Behavioral: General Parenting Education and Advice — Both the FAB group and the Control Group will receive routine family support services from collaborating NGOs, including education on managing the emotional and behavioral symptoms of children with NDD. To control for the interaction/social effect present in the FAB group, the Control Group will also receive four video-conferencing sessions guided by a trained research assistant over 12 weeks. These sessions will facilitate parents to discuss their parenting challenges, identify parenting traps, and provide general parenting advice as recommended by the Child Assessment Services, Department of Health under the HKSAR government.
  Arms: Control Group

SUMMARY:
The study aims to examine the effectiveness of a psychotherapy approach called Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB) in improving the psychological health of parents of young children with neurodevelopmental disorders (NDD) and reducing the emotional and behavioral symptoms of NDD children. The study will involve 154 Cantonese-speaking parents of children aged 2-6 years diagnosed with NDD in Hong Kong. The study hopes to find that FAB can improve parent-child dyads' health outcomes by enhancing psychological flexibility, parental psychological health, and mindful parenting skills.

DETAILED DESCRIPTION:
Background: Neurodevelopmental disorders (NDDs) are heterogeneous disorders that typically develop in early childhood and are characterised by developmental deficits that result in impaired personal, social, and/or occupational functioning. In Hong Kong, according to the latest statistical report from the Education Bureau, it is estimated that at least 71,320 preschool and school-age children have been diagnosed with NDD and are currently receiving special education and/or health care services. It is well documented that NDD children have less clear communication signals to their parents and poorer prosocial skills.

Continued failures and difficulties in understanding and responding to children's needs may prevent parents from developing positive parenting behaviours, which can negatively impact parents' psychology and ultimately snowballing their NDD child's emotional and behavioural symptoms. To our knowledge, effective interventions that specifically target the mental health of parents caring for young children with NDD to improve outcomes for both parents and children are extremely scarce. To address this study gap, this study will implement and examine the effectiveness of the Facilitator-guided Acceptance and Commitment Bibliotherapy, a facilitator-guided manual reading psychotherapy approach that explicitly targets the psychological needs of parents, in parents of young children with NDD in On-site Pre-school Rehabilitation Service (OPRS) teams.

Objectives: To examine the effectiveness of the Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB) and general parenting advice, in comparison to the control (general parenting advice only), on outcomes related to parental psychological health (parenting stress, symptoms of depression and anxiety, psychological flexibility), parenting behaviour, as well as the child's emotional and behavioural symptoms over 6 months of post-intervention period.

Hypotheses to be tested: Compared to the control group alone, FAB participation could achieve the following goals: reduce parents' parenting stress and NDD children's emotional and behavioural symptoms, reduce parental depressive and anxiety symptoms, improve psychological flexibility and nurturing behaviours of mindful parenting, and reduce the use of health care and rehabilitation services for young children with NDD over 6 months of post-intervention period.

Design: A multi-centre, two-arm randomised controlled trial (RCT) with a repeated-measures parallel-group design

Subjects: 154 Cantonese-speaking parents of children aged 2-6 years diagnosed with neurodevelopmental disorders

Instruments: Validated questionnaires

Interventions: Facilitator-guided Acceptance and Commitment Bibliotherapy (FAB)

Main outcome measures: parental psychological health outcomes and the child's emotional and behavioural symptoms

Data analysis: Generalised estimating equation analyses with covariates adjustments

Expected results: After participating in FAB, parents will become more psychologically flexible in caring for their children with NDD. Parents also acquire better psychological health and mindful parenting skills, leading to eventful improvements in parent-child dyads health outcomes.

ELIGIBILITY:
Parents of young children with NDD who fulfil the following criteria will be recruited:

* Cantonese-speaking Hong Kong residents,
* aged ≥ 21 years,
* have a child aged between two and six years old (preschool age) with a clinically documented diagnosis/suspected NDD diagnosis according to DSM-5 criteria (e.g., ASD, ADHD, developmental delay) and enrolled in the SWD subvented pre-school rehabilitation services offered by NGOs,
* caregivers who adopted the responsibility of taking care of the child, living together with the child, and
* have device(s) with internet access.

Parents of young children with NDD will be excluded if:

* has been diagnosed with severe mental illness(es),
* cognitive/language/communication/visual/hearing impairment(s) or disorders that may present difficulties in comprehending the content of the intervention; and/or
* are currently receiving another psychosocial, psychoeducational, or parenting intervention(s).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Parenting stress | Change from baseline assessment to immediate and 6 months post-intervention
  The Parenting Stress Index-Short Form (PSI-SF, 36 items, 5-point Likert scale). The PSI-SF evaluates parenting stress in three dimensions: parental distress, parent-child dysfunctional interaction, and difficult child behaviour (12 items each), with all items summed to indicate the total parenting stress [48]. Parents are asked to rate how much they agree or disagree with each statement using a 5-point Likert scale, ranging from "strongly agree" to "strongly disagree". Higher scores indicate higher levels of parenting stress. The Chinese version of PSI-SF (and its subscales) demonstrated strong convergent validity, discriminant validity and internal consistency (α =.79-.88) in Chinese parents.
Child's emotional and behavioural symptoms | Change from baseline assessment to immediate and 6 months post-intervention
  The Strengths and Difficulties Questionnaire (SDQ, 25 items, 3-point Likert scale). The SDQ consists of 25 items that assess five domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Each item is rated on a 3-point Likert scale, with higher scores indicating greater symptom severity for the emotional and behavioral problem domains and greater prosocial behavior for the prosocial behavior domain. The Chinese version of SDQ reported adequate test-retest reliabilities (ICC=.75-.86) and discriminant validity in Hong Kong parents.

SECONDARY OUTCOMES:
Parental symptoms of anxiety and depression | Change from baseline assessment to immediate and 6 months post-intervention
  The Hospital Anxiety and Depression Scale (HADS, 14-item, 4-point Likert Scale). The HADS is a widely used self-rating scale assessing symptoms of anxiety and depression (7 items per subscale). Each item is rated on a 4-point Likert scale, ranging from 0 to 3, with higher scores indicating greater symptom severity, and its total subscale score ≥ 8 indicates considerable symptoms. The total score for each subscale ranges from 0 to 21, with higher scores indicating more severe anxiety or depression symptoms. This Chinese version of HADS demonstrated adequate construct validity and internal consistency in the Hong Kong sample (α =.67-.79).
Parental psychological flexibility | Change from baseline assessment to immediate and 6 months post-intervention
  The Psyflex questionnaire (6-item, 5-point Likert scale). The Psyflex questionnaire consists of 6 items that use a 5-point Likert scale to assess different aspects of psychological flexibility, such as the ability to be present in the moment, to accept difficult thoughts and emotions, and to focus on what matters most. Higher scores on the Psyflex questionnaire indicate greater psychological flexibility, which has been associated with better mental health outcomes. The Psyflex possesses excellent convergent validity, divergent validity, and reliability (Raykov's r = .91). Its Chinese version has been validated in the PI's work.
Parenting behaviour | Change from baseline assessment to immediate and 6 months post-intervention
  is a self-report measure consisting of 31 items, which use a 5-point Likert scale to assess mindfulness in parenting. The questionnaire evaluates various aspects of mindfulness in parenting, such as being present with one's child and responding to their emotions with compassion. Parents are asked to rate how frequently they engage in each behavior, with responses ranging from "never" to "very often". The IM-P generates a total score, as well as scores for five subscales: "Listening with Full Attention", "Emotional Nonreactivity to Child Distress", "Nonjudgmental Acceptance of Parenting Experience", "Compassionate Responding to Child's Needs", and "Emotion Regulation in Parenting". Higher scores on the IM-P reflect greater levels of mindfulness in parenting. The Chinese version of IM-P, which has been used in our Co-I's trial, demonstrated good convergent validity and internal consistency (α =.70-.84) among parents.
Child's use of health care and rehabilitation services | Change from baseline assessment to immediate and 6 months post-intervention
  The types and frequencies of rehabilitation service use from private and/or public health sectors per month over the past six months will be reported by parents, and cross-checked with the records provided by the On-site Pre-school Rehabilitation Services (OPRS) teams.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Hong Kong Sheng Kung Hui Welfare Council Limited, Hong Kong
  - The Chinese University of Hong Kong, Shatin